CLINICAL TRIAL: NCT05140993
Title: The Role of Emotional and Orientation Support in Prevention of Postoperative Delirium Among Elderly Surgical Patients - a Multiple-crossover Clinical Trial
Brief Title: The Role of Emotional and Orientation Support in Prevention of Postoperative Delirium Among Elderly Surgical Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barak Cohen, MD (Other Government)
Responsible Party: Sponsor-Investigator, Barak Cohen, MD, Vice Chair Division of Anesthesiology, Intensive Care Medicine and Pain management, Tel-Aviv Medical Center, Sackler faculty of medicine, Tel-Aviv University, Israel, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 0483-21
Record Dates: First submitted 2021-09-29; First posted 2021-12-02 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: suggest a single-center, open-label, multiple-crossover trial in which all eligible patients will be enrolled, and the intervention (providing extended emotional and orientation support) will be altered every two weeks against the control, which is the current clinical practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- extended support (Experimental): providing extended emotional and orientation support
  Interventions: Behavioral: extended emotional and orientation support
- common practice (No Intervention): The hospital routine clinical standard- not providing extended emotional and orientation support

INTERVENTIONS:
Behavioral: extended emotional and orientation support — extended emotional and orientation support
  Arms: extended support

SUMMARY:
Postoperative delirium is common and associated with significant adverse outcomes. Its etiology is unknown, and little is known about associated risk factors. The investigatorea aim to test whether providing emotional and orientation support can reduce the risk of postoperative delirium in elderly patients undergoing elective non-cardiac surgery. Specifically, the investigators will test whether allowing such patients to keep their hearing and visual aids and be escorted into the operating room by a family member until anesthesia induction reduces the incidence of postoperative delirium. Delirium will be actively screened as part of our institution's clinical practice starting at PACU admission and for a minimum of 2 postoperative days. The investigators will use a multiple cross-over design to enroll all eligible patients and alternate between the intervention and our common practice (removing sensorial aids in the preoperative area and not allowing patients' escort beyond that point) every 2 weeks for up to 2 years.

DETAILED DESCRIPTION:
The world population is constantly growing older, and life expectancy in the western world is well over 80 years. The older population suffers more severe comorbidities, yet needs more surgical care. Anesthesiologists and surgeons are therefore required to care for older and sicker patients, often undergoing longer and more complex procedures than in the past.

Delirium is one of the most common adverse events experienced by hospitalized elderly patients. It is defined as an acute and fluctuating state characterized by altered awareness, behavior, emotional state, or thinking, and is associated with other morbidities as well as with mortality. Postoperative delirium (POD) affects between 10% and 50% of elderly surgical patients, depending on patients' baseline morbidities, the type of surgical procedure, and the tools and criteria used for diagnosis. POD is certainly the most common postoperative complication in this patient population, and is strongly associated with other postoperative adverse outcomes and mortality. Many societies and task-forces now recommend routine screening for cognitive decline and delirium in the perioperative period.

Several risk factors have been identified to be independently associated with POD, such as age, sex, and preoperative cognitive level. Nonetheless, most of the known risk factors are not modifiable, and little is known regarding interventions that can potentially decrease the risk of POD.

The division of Anesthesia and Intensive Care in the Tel-Aviv Medical Center has been conducting a quality improvement project since 2019, in which all surgical patients 70 years or older having elective non-cardiac non-cranial surgery are screened postoperatively for POD using the validated 4A's test starting in the post-anesthesia care unit (PACU) and for at least two postoperative days. The participants are also screened for preoperative cognitive decline, and monitored for other significant postoperative adverse events. Nearly 2000 eligible patients have been analyzed to date.

POD incidence in our institution is over 14%, and the investigators found a strong association between preoperative cognitive decline and POD, as also demonstrated by others. Interestingly, the investigators also demonstrated a strong association between delirium diagnosis in PACU and a later diagnosis in the surgical ward, suggesting that screening for delirium as early as PACU admission is important.

Many caregivers feel that the cognitive and emotional state in which patients are during induction of general anesthesia has a great impact on their immediate recovery. Frail and elderly patients are probably even more sensitive to this effect. Our common clinical routine while caring for adult surgical patients is to have a family member or friend escorting patients into the preoperative admission area, but not into the operating room. Similarly, our nursing practice includes the removal of hearing and visual aids prior to entry into the operating room. Since older patients are more prone to POD, the negative impact of separating them from their emotional and orientation support is presumably significant. In contrast, it is very common to have a family member escorting pediatric patients into the operating room and supporting them until anesthesia induction. The investigators previously conducted a pilot feasibility project in which the investigators allowed a family member of 50 elderly patients to escort them into the operating room. The investigators found that the process is feasible and simple. Moreover, all participants were satisfied and reported that they would be happy to use such an option in the future, and no family member was overwhelmed or had any adverse event as a consequence of entering the operating room.

The investigators therefore wish to test the hypothesis that allowing patients 70 years or older having non-cardiac non-cranial surgery to enter the operating room escorted by a supporting person and keeping their hearing and visual aids until anesthesia induction reduces the incidence of postoperative delirium during the initial two postoperative days.

Postoperative delirium is the most common postoperative complication in the elderly population, and has major impact on length of hospitalization, and postoperative morbidity and mortality. There are currently no known preventive interventions to reduce this risk. The investigators suggest a simple and safe logistic institutional intervention that can potentially reduce this risk.

Objectives

To test whether emotional and orientation support provided to surgical patients over 70 years of age reduces the incidence of postoperative delirium during the initial 2 postoperative days.

Research questions:

Are patients ≥ 70 years having non-cardiac non-cranial surgery who are being escorted into the operating room by a supporting person and keeping their hearing and visual aids, at reduced risk of postoperative delirium during the initial two postoperative days, compared to the clinical routine of separating patients from such emotional and orientation support before entry into the operating room?

Primary aim - to test the hypothesis that providing elderly surgical patients with emotional and orientation support until anesthesia induction reduces the risk of postoperative delirium, compared to the clinical routine of removing such support in the preoperative admission area.

Methods and Measurements

The investigators suggest a single-center, open-label, multiple-crossover trial in which all eligible patients will be enrolled, and the intervention (providing extended emotional and orientation support) will be altered every two weeks against the control, which is the current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 70 years
2. having non-cardiac and non-cranial surgery in the Tel-Aviv Medical Center

Exclusion Criteria:

1. Known psychiatric or severe neurologic disorder (e.g., Alzheimer's disease, past stroke)
2. Preoperative cognitive decline (MiniCog test result < 3 points)
3. Not planned to be extubated and awaken at surgery conclusion
4. Known inability to cooperate with postoperative delirium screening (language barrier, aphasia)

Ages: 70 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | Up to 30 postoperative days
  A composite outcome of postoperative delirium, consisting of at least of the following - a positive 4A's test, positive 3D-CAM test, or delirium symptoms described in the nursing notes.

CONTACTS AND LOCATIONS:
Overall Officials: Barak Cohen, MD, Principal Investigator — Tel-Aviv Medical Center, Sackler faculty of medicine, Tel-Aviv University, Israel
Locations (1):
- Division of Anesthesiology, Intensive Care Medicine and Pain management, Tel-Aviv Medical Center, Sackler faculty of medicine, Tel-Aviv University, Israel, Tel Aviv, Israel